CLINICAL TRIAL: NCT01631669
Title: Prophylaxis of Heterotopic Ossification (HO) in Wartime Extremity Injuries, a Randomized Clinical Trial
Brief Title: Celecoxib for Primary Prophylaxis of Combat-Related Heterotopic Ossification
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 352511; 110587 (Other: FDA IND)
Record Dates: First submitted 2012-06-27; First posted 2012-06-29 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Ossification, Heterotopic
Keywords: Ossification; Heterotopic Ossification
MeSH Terms: conditions — Ossification, Heterotopic | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Celebrex (Experimental): Receive Celebrex
  Interventions: Drug: Celecoxib
- Control (No Intervention): no placebo administered

INTERVENTIONS:
Drug: Celecoxib — 200 mg Q 12 hours orally
  Other Names: Celebrex
  Arms: Celebrex

SUMMARY:
Hypotheses:

H1: Celecoxib, when given less than five days after injury will result in a statistical decrease in the incidence and/or severity of radiographically apparent Heterotopic Ossification when compared to controls.

H2a: A biomarker profile will accurately predict which patients in the treatment group will respond to Celecoxib prophylaxis for Heterotopic Ossification.

H2b: A biomarker profile will accurately predict which patients in the control group are at highest risk of developing Heterotopic Ossification

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. ISS ≥9 (a traumatic trans-tibial amputation is an ISS of 9)
2. Extremity Wound ≥75cm2 requiring operative intervention
3. Minimal age of 18 years

Exclusion Criteria:

The following co-morbidities will result in exclusion from study:

1. Coronary Artery Disease,
2. Diabetes Mellitus (IDDM or T2DM),
3. Peripheral Vascular Disease,
4. Age >65,
5. Connective tissue disorders,
6. Immunosuppression,
7. Clinically-evident peptic ulcer disease,
8. Substantial renal dysfunction (as assessed by a serum creatinine >1.5 or calculated creatinine clearance of <50),
9. Spine-injured patients who have recently received or are going to receive spinal fusion as determined by the evaluating neurosurgeon or orthopaedic spine surgeon at LRMC,
10. Severe penetrating or hemorrhagic traumatic brain injury,
11. Endoscopic gastrointestinal interventions,
12. Pregnancy or women of childbearing who does not take a pregnancy test and effective method of birth control.
13. Known hypersensitivity to Celebrex, Aspirin, other NSAIDs, or Sulfonamides.
14. History od Asthma, Urticaria, or allergic-type reactions after taking Aspirin or other NSAIDs.
15. Hepatic Impairment
16. Warfarin
17. Lithium
18. Drugs known to inhibit CYP2C9 Liver Enzymes
19. Subjects known or suspected to be poor CYP2C9 metabolizers
20. Concomitant use with ACE Inhibitors and Angiotension II Antagonists

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Prophylaxis of Heterotopic Ossification (HO) in Wartime Extremity Injuries, a Randomized Clinical Trial | 3 years
  Incidence and severity of HO

SECONDARY OUTCOMES:
Prophylaxis of Heterotopic Ossification (HO) in Wartime Extremity Injuries, a Randomized Clinical Trial | 3 years
  1. Overall rate of impaired wound healing.
  2. Overall time to fracture union (if applicable)
  3. Overall rate of nonunions (if applicable)
  4. Overall rate of drug-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Forsberg, MD, Principal Investigator — Walter Reed National Military Medical Center
Locations (2):
- Walter Reen National Military Medical Center Bethesda, Bethesda, Maryland, United States
- Landstuhl Military Medical Center, Landstuhl, Germany

REFERENCES:
- [Background] Forsberg JA, Pepek JM, Wagner S, Wilson K, Flint J, Andersen RC, Tadaki D, Gage FA, Stojadinovic A, Elster EA. Heterotopic ossification in high-energy wartime extremity injuries: prevalence and risk factors. J Bone Joint Surg Am. 2009 May;91(5):1084-91. doi: 10.2106/JBJS.H.00792. PMID 19411456
- [Background] Potter BK, Burns TC, Lacap AP, Granville RR, Gajewski DA. Heterotopic ossification following traumatic and combat-related amputations. Prevalence, risk factors, and preliminary results of excision. J Bone Joint Surg Am. 2007 Mar;89(3):476-86. doi: 10.2106/JBJS.F.00412. PMID 17332095